CLINICAL TRIAL: NCT05620069
Title: The Effect of Listening to Music on Sleep Disturbances in Patients With Acquired Brain Injuries
Brief Title: Music Listening and Sleep in Rehabilitation of People With Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejlefjord Rehabilitation (Other)
Collaborators: University of Aarhus (Other); Aalborg University (Other)
Responsible Party: Principal Investigator, Mette Underbjerg, Head of Research and Development, Vejlefjord Rehabilitation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2019-01-31; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Brain Injuries; Sleep Disturbance
Keywords: Brain injury; Acquired brain injury; Sleep disturbance; Music; Music therapy
MeSH Terms: conditions — Brain Injuries; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music listening at bed time (Experimental)
  Interventions: Other: Music listening
- Treatment as usual (No Intervention)

INTERVENTIONS:
Other: Music listening — Participants are asked to select one of four music playlists and listen to it for appr. 30 minutes at bedtime during the intervention period.
  Arms: Music listening at bed time

SUMMARY:
An Injury to the brain may lead to sleep-wake disturbances which may negatively influence functional recovery, quality of life and general rehabilitation.

The purpose of this study is to investigate the effect of music listening on sleep disturbances after acquired brain injury (ABI).

During a 2 week intervention period patients with ABI will listen to music for appr. 30 minutes before going to sleep. Records of their sleep quality are compared to records of sleep quality from 2 weeks without music intervention.

H1 Hypothesis: Music listening (ML) improves sleep quality after ABI in patients.

H0 Hypothesis: Music listening (ML) has no effect on sleep quality after ABI in patients.

DETAILED DESCRIPTION:
Participants are recruited from Vejlefjord Rehabilitation - a neurorehabilitation center in Denmark.

Patients who meet the inclusion criteria are enrolled in the study after informed consent. Participants are randomly allocated to two conditions (ML+Treatment as usual (TAU) or TAU only in a crossover design. Randomization is done by sealed envelope, and after two weeks of either ML+TAU or TAU the participants switch condition.

Participants are asked to select one of four music playlists and listen to it for appr. 30 minutes at bedtime during the intervention period. Participants will rate sleep quality and liking of the intervention.

Information about injury, demographic and socioeconomic status are derived from patient journals.

ELIGIBILITY:
Inclusion Criteria:

* in-patients with ABI being treated at Vejlefjord Rehabilitation during the entire project period
* age > 18 years
* sleep-wake disturbances corresponding a score of 5 or more on Pittsburgh Sleep Quality Index (PSQI).
* Mentally and physically capable of administering music equipment, actigraph and self-report questionnaires.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Change from baseline to after the 14-days intervention period
  Measured with the Pittsburgh Sleep Quality Index, range 0-21 with higher scores indicating more sleep problems.
Objective sleep quality | Change from baseline to after the 14-days intervention period
  Measured with wrist-worn actigraphy registrering body movements from which you can derive the sleep-wake pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Underbjerg, PhD, Principal Investigator — Vejlefjord Rehabilitation
Locations (1):
- Vejlefjord Rehabilitation, Stouby, Denmark

IPD SHARING:
Plan to Share IPD: No